CLINICAL TRIAL: NCT06340932
Title: Impact of Opioid Avoidance Protocol for ACL Reconstruction Surgery
Brief Title: Impact of Opioid Avoidance Protocol for ACL Reconstruction
Status: Completed | Type: Observational
Sponsor: Matthew Varacallo (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor-Investigator, Matthew Varacallo, Orthopedic Surgeon, Penn Highlands Hospital Duboia
Organization: Penn Highlands Hospital Duboia (Other)
Other Study IDs: CRS-119 (Pro00077191)
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: ACL Tear; Post Operative Pain
Keywords: Iovera; Cryoneurolysis; Multi-modal analgesics
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain, Postoperative | interventions — Celecoxib; Acetaminophen; Oxycodone; Tramadol; Bupivacaine; Capsules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Standard of Care: Treatment of pain as per standard of care. Patients will receive regional anesthesia blocks, acetaminophen, and as needed opioids; tramadol and oxycodone postoperatively for pain management.
  Interventions: Drug: Oxycodone; Drug: Tramadol; Drug: Bupivacaine Hydrochloride; Drug: Acetaminophen 500Mg Cap
- Opioid Avoidance: Preoperatively patients will receive cryoneurolysis of 5 sensory nerves that innervate the knee 7 to 21 days before surgery. Patients will receive perioperative NSAIDs and acetaminophen along with regional anesthesia. For postoperative pain control patients will receive scheduled acetaminophen and NSAIDs and may request opioids as needed.
  Interventions: Device: Iovera; Drug: Celecoxib; Drug: Acetaminophen; Drug: Oxycodone; Drug: Tramadol; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Device: Iovera — Cryoneurolysis of 5 sensory nerves (Intermediate branch of the AFCN, Medial Femoral Cutaneous Nerve, Suprapatellar branch of the saphenous nerve, 2 branches of the infrapatellar branch of the saphenous nerve) causing Wallerian degeneration
  Groups: Opioid Avoidance
Drug: Celecoxib — 200mg BID
  Other Names: Celebrex
  Groups: Opioid Avoidance
Drug: Acetaminophen — 1000mg q8h
  Other Names: Tylenol
  Groups: Opioid Avoidance
Drug: Oxycodone — As needed
Drug: Tramadol — As needed
Drug: Bupivacaine Hydrochloride — 20mL of 0.25% bupivacaine HCl adductor canal block and 15mL of 0.25% bupivacaine HCl (+/- 5mL of normal saline) iPACK
Drug: Acetaminophen 500Mg Cap — 500mg q6h prn
  Groups: Standard of Care

SUMMARY:
This is a prospective, quasi-experimental, cohort study comparing patients treated with one of two postoperative pain management protocols. The two protocols assessed will be the current standard of care protocol for Anterior Cruciate Ligament Reconstruction (ACLR) postoperative pain control utilized by Dr. Matthew Varacallo and then an opioid avoidance protocol that is planned to be implemented on the Spring of 2024. The study is voluntary, however all patients will be treated with either of the two protocols depending on their date of surgery. This study will include patients aged 15 years and older who consent to the participation in the study. Patients will be identified utilizing the operative surgeon's appointment calendar and will be screened and offered inclusion in the study if applicable at their pre-operative visit. Data will be collected via patient medication and pain diary, phone call, and clinician administration of standardized outcome questionnaires. Patients will be included in the standard of care group if ACLR is performed prior to the change in protocol in the Spring of 2024 or the opioid avoidance group if performed after the protocol change.

The primary objective of this study is to evaluate the effect of the opioid avoidance protocol on opioid use in milligrams of morphine equivalent (MME) from postoperative day (POD) 0 to 7 after ACLR compared to the current standard of care pain management protocol.

Secondary objectives are to:

* evaluate the effects of an opioid avoidance protocol on the daily average numeric rating scale (NRS) pain scores from POD0-7
* evaluate the effects of an opioid avoidance protocol on the daily worst NRS pain score from POD0-7
* evaluate the ability to recover opioid free through 7, 30, and 60 days
* evaluate the quality of recovery 15 (QoR-15) scores on POD2
* assess the number of opioid prescriptions required by patients in the 60 day recover period
* assess Knee Injury and Osteoarthritis Outcome Score (KOOS) pain and symptom scales at 8 weeks post-operatively between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15 years or older at screening.
* Primary diagnosis of ACL injury as evidenced by MRI or similar imaging study and are scheduled to undergo ACLR with or without meniscal repair/meniscectomy
* Non-pregnant patients with verbal confirmation that they are not planning to become pregnant during the study period.

  i. Female subjects must have a confirmatory negative pregnancy test as part of the routine pre-operative laboratory testing ii. Subjects must endorse a plan to utilize contraceptives (condoms, hormonal birth control, IUD, etc.) for any sexual activity during the study period.
* English speaking patients
* Provision of informed consent with ability to adhere to the study visit schedule and complete all study assessments.

Exclusion Criteria:

* Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications
* History of contralateral ACL repair within 1 year of screening
* Multi-ligament injury requiring reconstruction
* Inability to return to the study doctor's clinic for postoperative visits
* Pregnant or trying to become pregnant
* Breastfeeding
* Have a severe chronic pain condition that in the opinion of the study doctor may impact post-surgical outcomes of analgesic and opioid usage (i.e., fibromyalgia, cancer, sickle cell disease)
* Have a known contraindication to the iovera° device, including any of the following:

  i. Cryoglobulinemia (presence of abnormal proteins in the blood that thicken in cold temperatures) ii. Paroxysmal cold hemoglobinuria (an autoimmune disorder where cold-reacting antibodies that attack and destroy red blood cells) iii. Cold urticaria (temporary itchy welts [hives] on skin exposed to cold temperatures) iv. Raynaud's disease (which causes some areas of the body, such as fingers and toes, to feel numb and cold in response to cold temperatures) v. Open and/or infected wounds at or near the study treatment site vi. Coagulopathy (problems with blood clotting)
* Have poorly controlled mental illness that in the opinion of the study doctor may meaningfully impact study treatment outcomes, including any of the following:

  i. Mood disorder (for example, major depression, bipolar) ii. Psychotic disorder (for example, schizophrenia)
* Have a history, suspicion, or clinical manifestation of:

  i. Alcohol abuse or dependence ii. Illicit drug use iii. Opioid abuse or dependence (greater than or equal to 40 mg morphine equivalent dose by mouth per day in the past 30 days)
* Pregnant or planning to become pregnant during the study period

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents (15 years of age or older) or Adults undergoing primary ACL reconstruction with or without meniscal repair.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-04-27 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumption from post-operative day 0 to 7 | 7 days
  Total use of opioids in milligrams of morphine equivalent from day 0 through day 7

SECONDARY OUTCOMES:
Average daily pain score via numeric rating scale (NRS) | 7 Days
  Average daily pain each day from POD0-7
Average daily worst pain score via NRS | 7 days
  Average of highest pain scores daily
Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Subscale Score | Week 8
  Pain subscale of the KOOS questionnaire
Quality of Recovery-15 | Day 2
  QoR15 score on POD2
Pittsburgh Rehabilitation Participation Scale Score | 8 weeks
  Ability to participate in physical therapy weekly
KOOS symptom subscale score | Week 8
  Symptom subscale of the KOOS questionnaire
Quantity of opioid prescriptions utilized at day 30 and 60 | Day 30 and Day 60
  Number of opioid prescriptions filled by patient at day 30 and 60
Opioid-free at day 7, day 30, and day 60 | Days 7, 30, and 60
  Percentage of patients who did not utilize opioid prescriptions at 3 time points

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Highlands Dubois, DuBois, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No